CLINICAL TRIAL: NCT06159218
Title: Eosinophil Associated Proteins and Microbiome Profiling in Adults With Eosinophilic Oesophagitis at a Single UK Tertiary Centre
Brief Title: Eosinophilic Oesophagitis Assessment With String Testing
Acronym: EoEAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021.0276; IRAS (Other: 303427)
Record Dates: First submitted 2022-11-24; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: Adult patients with Eosinophilic Oesophagitis will undergo a swallowed string test just prior to their scheduled endoscopy. No additional endoscopy will be requested than as per routine care. String test will be analysed for biomarkers and the microbiome to compare against disease severity and medical therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole (Active Comparator): Patients with active EoE who have been started on omeprazole as treatment
  Interventions: Device: CEST - coiled oesophageal string test
- Budesonide (Active Comparator): Patients with active EoE who have been started on budesonide as treatment
  Interventions: Device: CEST - coiled oesophageal string test

INTERVENTIONS:
Device: CEST - coiled oesophageal string test — All patients will swallow a small string (CEST) which will be removed and then analysed for biomarkers and microbiome.

SUMMARY:
Eosinophilic oesophagitis (EoE) is an inflammatory condition of the oesophagus (food pipe) that can lead to difficulty swallowing and to food to getting stuck and has become increasingly common over the past 40 years.

EoE is triggered by a protein in the diet but alterations to the types of bacteria (microbiome) in the oesophagus may also be involved. EoE is diagnosed with gastroscopy (a thin camera test via the mouth) where 6 tiny samples (biopsies) are taken. Treatment is either with removing food groups from the diet or medications including steroids (budesonide) or a proton pump inhibitor (PPI, omeprazole). The aim is to improve symptoms and to stop scar tissue forming that can cause food to get stuck.

Patients with EoE will need to undergo many gastroscopies over their life, which even with sedation can be a daunting experience. There has been research into less invasive tests and two previous studies have shown that a thin swallowed string may be able to detect substances (biomarkers) that indicate how severe the EoE is. These studies were small and it is not known how the biomarkers change with different treatments or how well they relate to symptoms and findings with endoscopy.

In this study the investigators will ask adults with EoE to swallow a thin string made of rayon for 30 minutes, with one end taped to the cheek, which the investigators will analyse for biomarkers and bacteria, on the same day as their routine gastroscopy and also perform a symptom survey. The investigators will also take an extra 2 biopsies to analyse the nerves which may explain why some patients have more symptoms than others. The investigators will repeat the string test on their next endoscopy, to assess what the changes have been in response to their treatments. These findings may improve understanding on how to monitor EoE in less invasive ways in future.

DETAILED DESCRIPTION:
Eosinophilic oesophagitis (EoE) is a chronic progressive inflammatory condition of the oesophagus first described in 1978 but not recognised as distinct diagnosis until 1993, affecting both children and adults. It is characterised by eosinophilic infiltration of the oesophageal epithelium and can lead to difficulty swallowing, oesophageal strictures, food bolus obstruction, and symptoms mimicking gastro-oesophageal reflux disease (GORD). 23% adults with dysphagia and 50% with food bolus obstruction are diagnosed with EoE, meaning it is a common condition encountered by Gastroenterologists. Recent systematic reviews have estimated that EoE has a pooled prevalence of 28-34 per 100,000 population, but the incidence has risen remarkably over the past four decades.

EoE can occur at any age, with a rising incidence in children and adults aged 30-50 years and studies have shown that it can significantly impact on health related quality of life by impairing social and psychological functioning. It is more common in males and in those with allergic conditions such as asthma, eczema and rhinitis, suggesting a food or aeroallergen trigger. Diagnosis is obtained by gastroscopy with a minimum of six oesophageal biopsies recommended by international guidelines, due to its potentially patchy distribution. Hallmark endoscopic appearances of the oesophagus have been described and include oesophageal rings, longitudinal furrows, oedema, exudate, and narrowing. Oesophageal biopsies must show > 15 eosinophils (eos) per high powered field (HPF) infiltrating the oesophageal mucosa, as to not be mistaken with other conditions such as GORD which may also exhibit eosinophilic infiltration but at lower numbers. Other histological features include eosinophil micro-abscesses, basal zone hyperplasia, dilated intercellular spaces, eosinophil surface layering, papillary elongation and lamina propria fibrosis.

Once a diagnosis has been made, treatment of EoE is with food elimination diets, proton pump inhibitors (PPI), or topical glucocorticoids, such as budesonide orodispersible tablet (BOT). In a small subgroup of patients, immunomodulatory drugs such as azathioprine or 6-mercaptopurine might be required, and research is ongoing into monoclonal antibody therapy. The aim of treatment, as described in recent European and American Gastroenterological Association (AGA) and Joint Task Force on Allergy Immunology Practice Parameters (JTF) guidelines, is to alleviate symptoms, prevent stricture formation and achieve histological remission with < 15 eos/HPF infiltration.

Previous studies have shown that PPI may induce remission in 42% patients. Budesonide orodispersible table (BOT) may induce remission in 85% patients, but can be associated with the side effect of candidiasis in up to 10% patients. An empiric 6-food (dairy, wheat, soy, eggs, nuts, and seafood/shellfish) elimination diet induces histological remission in around 75% of patients, whereas a 4-food elimination diet (dairy, wheat, soy, and egg) induced histological remission in around 50% patients, and a 2-food elimination diet (dairy and wheat) may be effective for 40% patients. Elemental diet (amino acids) induces histological remission in 90% of patients but is impractical and only recommended for consideration after failure of medical therapy or elimination diets. Prolonged avoidance of dietary triggers may lead to drug-free sustained clinical and histological remission. Once a stricture has developed then endoscopic balloon dilatation may be required and can improve dysphagia in up to 75% of adults with oesophageal strictures, and is relatively safe with a perforation rate of only 1%, but has no effect on the underlying inflammatory process.

Systematic review with meta-analysis found no statistical difference between PPI and BOT, however there are few head to head studies comparing the treatments and long term evidence for BOT is still lacking; indicating the need for further prospective studies. European guidelines therefore currently do not favour one treatment over another and state that the choice of therapy should be individually discussed with the patient and may be interchangeable over time. Treatment effectiveness should be assessed with repeat gastroscopy with oesophageal biopsies after 6-12 weeks.

Gastroscopy involves placing a thin flexible camera into a patient's mouth and advancing it to the oesophagus, stomach and duodenum. The procedure takes approximately 5 minutes, during which biopsy forceps are placed through a 2.8mm channel on the standard gastroscope to obtain oesophageal mucosal biopsies for histological analysis. Although topical anaesthetic may be applied to the back of the throat and intravenous sedation given, for many patients, gastroscopy remains an unpleasant and daunting experience. Transnasal endoscopy (TNE) has more recently been developed and potentially offers patients a more comfortable procedure due to the reduced diameter of the gastroscope, but due to the need for lifelong surveillance, there has been a move for even less invasive and less costly methods.

The GI string test (EnteroTestTM) was first developed in 1970 for sampling microorganisms from the small intestine. The original test involved swallowing a small, weighted gelatin capsule to which a string was attached and the other end taped to the patients cheek. The capsule reaches the duodenum where it detaches and is excreted naturally and the string left in situ overnight. The string is then pulled out via the mouth and can be analysed. Over the years it has been used to analyse biliary composition, culture intestinal tuberculosis, and profile the distinct microbiome in the oesophagus using 16S rRNA gene sequencing, as accurately as with mucosal biopsy.

The potential for oesophageal string testing (EST) to monitor EoE activity has been suggested by a previous study using an overnight swallowed string test in 41 children correlated with EoE activity on biopsy, which could distinguish between active EoE, treated EoE, GORD and normal oesophagus, using measured ESGP (eosinophil secondary granule proteins) - including major basic protein 1 (MBP1), esosinophil peroxidase (EPX), eosinophil derived neurotoxin (EDN) and eosinophil cationic protein (ECP). Also measured was the Chacot-Leyden crystal protein/galectin-10 (CLC/Gal-10), which is a primary cytosolic protein but is also present in the eosinophil's primary (coreless) granule. Each granule-associated protein carries different biochemical and functional properties relevant to proposed pathogenic mechanisms for oesophageal dysfunction and remodelling in EoE. These biomarkers were found to be elevated uniquely in active EoE, compared to treated EoE, GORD and normal controls.

Another previous study performed a one hour string test on 134 people with EoE or healthy control, comparing levels of eosinophil associated protein (EAP) including eotaxin-2 (Eot2), eotaxin-3 (Eot3), and MBP on EST to mucosal biopsy. Ackerman showed that these EST-captured eosinophil-associated biomarkers were proportionate on EST and mucosal biopsy levels, and also correlated with EoE activity as defined by mucosal eosinophil counts. These proteins on EST therefore had excellent sensitivity and specificity for identifying active EoE. They also surveyed patients, and 92% adults preferred the EST over gastroscopy to monitor their EoE.

Whilst these studies have shown the potential of intraluminal oesophageal biomarkers to reflect EoE activity, additional research is required to further characterise their relation to disease activity, correlation with symptoms and response to different treatments, which has not yet been described in the literature. This knowledge may improve our understanding of the pathogenesis of EoE and lead to new therapeutic targets in future, as well as reduce the need for surveillance endoscopy in EoE, which would be safer and more convenient for patients, and offer cost savings for healthcare resources.

The role of the microbiome is increasingly been appreciated in the development of immune mediated disease such as EoE, yet to date there are only a handful of studies on the oesophageal microbiome, finding distinct changes in EoE compared to GORD, adenocarcinoma and healthy patients. Further research in this area would be interesting to establish if the microbiome is different in active EoE vs remission, and how this may affect disease severity and symptoms, which again may lead to new therapeutic targets in future.

In addition, it is not known whether people with EoE have altered sensitivity in their oesophagus as part of the remodelling from the chronic inflammatory process. If sensation is increased this could lead to increased symptoms and if it is reduced then this coud lead to undiagnosed conditions including strictures and GORD. The calcitonin gene related peptide has recently been shown to be a marker of oesophageal sensory nerves, and has been shown to be closer to the oesophageal lumen in oesophageal hypersensitivity, however its relation to EoE has not yet been examined.

In this study the investigators will sample oesophageal biomarkers and the microbiome from adults with EoE, using a 30 minute string test, which will be performed on the same day as their routine gastroscopy an addition to validated symptom questionnaires. The investigators will repeat the string test after treatment courses with PPI, budesonide or dietary elimination, alongside their routine gastroscopy. During their gastroscopy the investigators will also take biopsies to check for the density and positioning of CGRP, to see if this is different in active and inactive EoE. The aim is to correlate biomarkers, CGRP and microbiome with endoscopic EoE activity and symptoms, to assess for changes in response to different treatments. and again may provide further insight into disease pathogenesis and lead to new therapeutic targets in future.

ELIGIBILITY:
Inclusion Criteria:

* Patient under the care of St George's University Hospital NHS Foundation Trust, London
* Diagnosis of EoE as defined by endoscopy with mucosal biopsy showing >15 eos/HPF
* Male or Female
* Age 18 to 90

Exclusion Criteria:

* Patients < 18 years old or >90 years old
* Patients with significant medical co-morbidities
* Patients unable to provide consent for study participation
* Patients who have had complications from their endoscopy or EoE treatment
* Patients who have previously undergone oesophageal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Do eosinophil associated protein (EAP) biomarkers detected with string testing correlate with peak eosinophil count (eos/HPF) on endoscopic mucosal biopsy in adults with eosinophilic oesophagitis (EoE)? | 12 weeks
  Measurement of string biomarker levels in comparison to mucosal eosinophil counts
How does the oesophageal microbiome, sampled with string testing, change after treatment for EoE? | 12 weeks
  Measurement of bacterial abundance (sequences per sample) on string testing
How does the density of calcitonin gene related peptide (CGRP) in the oesophageal mucosal biopsy change after treatment for EoE? | 12 weeks
  Assessment of change in density of CGRP in mucosa after treatment for EoE

SECONDARY OUTCOMES:
How do EAP detected with string testing change in response to treatments for EoE? | 12 weeks
  Comparison of string biomarker levels in those on omeprazole vs budesonide therapy
How does the oesophageal microbiome, sampled with string testing differ in EoE treatments? | 12 weeeks
  Comparison of bacterial abundance (sequences per sample) on string testing in those on omeprazole vs budesonide therapy

CONTACTS AND LOCATIONS:
Locations (1):
- St Georges University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No